CLINICAL TRIAL: NCT02693561
Title: Effectiveness of Deep Breathing, a Self-Help Book and Additive Effects of The Two Interventions in Cigarette Consumption, Anxiety and Depression and Motivation to Stop Smoking in Students of the Anhembi Morumbi University
Brief Title: Effects of Deep Breathing,Self-Help Book in Cigarette Consumption,Anxiety,Depression and Motivation to Stop Smoking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhembi Morumbi University (Other)
Responsible Party: Principal Investigator, Iris Galdino Ueda, Principal Investigator, Anhembi Morumbi University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AnhembiMU
Record Dates: First submitted 2016-02-10; First posted 2016-02-26 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Smoking Cessation
Keywords: Self-help book; Deep breathing
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Deep Breathing Exercises (Active Comparator): Technical Deep Breathing.
  Interventions: Behavioral: Deep Breathing Exercises
- Self-Help Book (Active Comparator): Reading the self-help book.
  Interventions: Behavioral: Self-Help Book
- Deep Breathing Exercises and Book (Active Comparator): Technical Deep Breathing and Reading the self-help book.
  Reading the self-help book and will be trained by the physical therapist to perform deep breathing.
  Interventions: Behavioral: Deep Breathing Exercises
- Control (No Intervention): Not suffer any intervention

INTERVENTIONS:
Behavioral: Deep Breathing Exercises — Technical Deep Breathing: Deep breathing is to deep breath and slowly through the nostrils until total lung capacity. At the end of inspiration is kept a few seconds of apnea and started after the expiration slowly. End-expiratory apnea will remain a few seconds to start new inspiration cycle. With this process the individual breathe about 6 times per minute. Breath learning occurs through visual feedback. In the intervention group will be held deep breathing for 10 minutes. Subjects will be instructed to deep breath for 10 minutes 2 times a day for 15 days beyond the period in which they cleft, which is one of the symptoms of withdrawal syndrome. Control and frequency of deep breathing will be obtained weekly through specific daily fill, which will be provided weekly.
  Arms: Deep Breathing Exercises; Deep Breathing Exercises and Book
Behavioral: Self-Help Book — Reading the self-help book.
  Arms: Self-Help Book

SUMMARY:
Smoking is an important public health issue. The self help books may have important motivational implications which associated with deep breath exercises could cease the habit. Goals: Verify the effectiveness of the deep breaths exercises from the self help books along with the two motivational interventions to quit smoking on the anxiety, depression and daily consumption levels. Method: The study will be both prospective and controlled. Individuals will be distributed randomly in 4 different groups: The first group will be doing the deep breath exercises, the second group will read a self help book, the third group will do both reading and exercises and the fourth group will be the control. Anxiety, depression, motivational level and the cigarettes daily consumption will be evaluated previously and after the 15 days intervention. Expected results: Decreasing in anxiety, depression and cigarette consumption plus an increase in the motivation to quit smoking.

DETAILED DESCRIPTION:
Smoking is a major public health problem. According to the WHO (World health organization) it's considered a pandemic issue which kills around 5 million people from related diseases.

This is a growing problem in all South American countries specially where poverty and the lack of instruction make people more vulnerable to the addiction. In addition, the smoking habit has been integrated to these countries cultures because of their economical dependence of it and ostensive marketing.

However, nowadays smoking harm effects are well known including the high risk of developing COPD (chronic obstructive pulmonary disease), heart diseases and many other forms of neoplasms.

The problems concerning smoking were first documented 40 years ago and are still one of the major causes of death which could be prevented. The medical costs associated with its treatment go far beyond the economical benefits from producing and commercializing tobacco.

It's estimated that in 2025, there will be 10 million people dying from tobacco consumption if the world panorama stays as it is. 90% of the teenagers who starts smoking become addicted by they are 19 years old.

According to the Smoking cessation guidelines - 2008 to stop smoking the addiction is recognized as a chronic condition and the interventions to change habits tends to be repeated as it's hard to get a efficient treatment. Even though, the stop smoking is associated in an increase of life quality and that's why it should be stimulated.

Three main mechanisms influence smoking, the first one is positive reinforcement, which is related to the release of acetylcholine, norepinephrine, serotonin, and GABA in the nervous central system caused by the action of nicotine that reduces appetite, improves mood and concentration and generate feelings of pleasure. The second is negative reinforcement, which generates the maintenance of cigarette use to prevent the symptoms of withdrawal symptoms like anxiety, increased appetite, dysphoria, irritability and difficulty in concentrating. The third is the respondent conditioning, which is stimulated by environmental factors, negative emotions and positive that lead to the act of smoke. Thus smoking is a complex behavior that is related to lifestyle, while trying to quit smoking many individuals experience symptoms of withdrawal syndrome which is a major cause of relapse. Deep breathing technique is cited by smokers as a strategy to alleviate these symptoms abstinence.

Mcclernon et al. They found results suggesting that guided deep breathing exercises relieve the symptoms of abstinence nicotine.

According to Tharion et al. deep breathing decreases respiratory rate and increase the variability of heart rate, stimulates the autonomic parasympathetic nervous system and increase the relaxing substances such as endorphins, so it is recommended as a relaxation technique, as well as decreasing tension, anger and depression.

Initially, in addition to clinical assessment of the smoker and assessing the degree of dependence, to assess the degree of motivation is fundamental to start therapy approach.

Prochaska and Diclemente described a stage of readiness model for change (motivation), with the steps of pre-contemplation, contemplation, preparation, action and maintenance (prevent the return behavior, undertaking measures to prevent relapse). First described as a linear model and later as a spiral model, since patients often have relapses, and remain long periods in maintenance stage.

Thus, motivational interventions are critical in smoker's approach in all clinical situations, even when participants need medical support. The self-help books can be effective and have important implications for public health. These psycho-educational interventions are complex and usually contains multiple components that interact and involve behavioral changes of people.

Self-help materials, according to Song et.al., can be effective and less costly than individual therapy or group sessions, which for many people is hard to get. Currently there are materials available in audio, video and computer programs, though the writings are the most commons.

A literature review by Boyce et al. And published by the Cochrane Library, concluded that materials that are tailored individually, eg for pregnant women or young, are more effective than non-adapted materials and both are effective for smoking cessation compared to individuals who did not use the self help material.

In this review, there was no additional benefit of evidence of the use of self-help material associated with other interventions such as advice from a health professional or replacement therapy nicotine and no selected study in the review used the deep breathing technique associated with reading self help material.

However, such evidence is tested in developed countries and more research is needed to investigate its effects in countries where support to smokers are not easily available.

Polonio I.B et al. , Published in 2013 a self-help book with smokers auxiliary order containing the principles of behavioral intervention conducted on Santa Casa de Sao Paulo smoking clinic.

Finally, the hypothesis of the study is that the book will be an effective tool to reduce anxiety, depression and increased motivation to quit smoking, the investigators believe that the addition of deep breathing to read the book will enhance these effects.

ELIGIBILITY:
Inclusion Criteria:

* students from the Anhembi Morumbi University.
* minimum age of 18 years.

Exclusion Criteria:

* serious chronic diseases
* use of beta blockers.
* pregnant women.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Motivation measured with the Portuguese version of the "URICA" (Scale University of Rhode Island Change Assessment) | 2 weeks
  Scale developed by Prochaska and DiClemente, translated and validated to Portuguese used to measure the motivation to change. Determines different motivational stages in solving a problem. To classify the individual in the pre-contemplation stage (stage where the person does not consider the need for help), contemplation stage (the individual is aware of the problem), preparation stage (construction of attempts to change their behavioraction stage (taking concrete attempts to modify their behavior) and maintenance stage (the lifestyle is modified). The answers are given on a scale of 1 (completely disagree with the statement) to 5 (strongly agree). Each statement is linked to a different motivational stage and at the end of test, the investigators can determine which is the patient motivational level considering which stage his score was higher.

SECONDARY OUTCOMES:
Nicotine addiction measured whit the Portuguese version of the Fagerstrom test | 2 weeks
  Developed by Karl-Olov Fagerstrom, translated and validated for the Portuguese to be aware related to biochemical index enabling the classification of nicotine addiction as mild, moderate and severe. It consists of six items that help to estimate the degree of nicotine dependence. Each item features a score from 0 to 3 according to the response and the sum of the scores of the alternatives chosen classifies the degree of dependence. The total less than 2 points classifies a very low level of dependence, from 3 to 4 points classifies the low degree of dependence, 5 points classifies the average degree of dependence, 6 to 7 point classifies the high degree of dependence 8 to 10 points ranks very high degree of dependence.
Depression measured with the portuguese version of the "BDI" ( The Beck Depression Inventory). | 2 weeks
  Self-assessment measure of depression developed by Beck translated to Portuguese and validity. Consists of 21 items, including symptoms and attitudes, each with four alternatives with intensity going from 0 to 3.The items refer to sadness, pessimism, sense of failure, lack of satisfaction, guilty, sense of punishment, self-deprecation, self-accusations, suicidal ideas, crying spells, irritability, social withdrawal, indecisiveness, body image distortion, inhibition to work, sleep disturbance, fatigue, loss of appetite, weight loss, somatic concern. To evaluate and rank, according to the symptoms presented last week, the state of depression according to the sum of the scores of the chosen alternative. Total <10 points (without depression); 10-18 (mild to moderate depression); 19-29 (moderate to severe depression) and 30-63 (severe depression).
Anxiety measured with the Portuguese version of the "BAI" ( The Beck Anxiety Inventory) | 2 weeks
  Scale developed by Beck, translated and validated to Portuguese. It consists of 21 items that measure anxiety. The subject must answer how bothered he is with anxiety symptoms during the last week. The criteria for correction of scores constitute a scale of 0 to 3 points for each symptom (absolutely no = 0; 1 = slightly, moderately = 2; seriously = 3). The sum of the scores can range from 0 to 63 points. Therefore, the results differ in the degree of anxiety: minimum 0-10; mild-11-9; moderate level of 20 to 30 and severe level 31-63.

CONTACTS AND LOCATIONS:
Overall Officials: Iris Ueda, Principal Investigator — Anhembi Morumbi University; Igor Polonio, Study Director — Anhembi Morumbi University
Locations (1):
- Anhembi Morumbi University, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Muller F, Wehbe L. Smoking and smoking cessation in Latin America: a review of the current situation and available treatments. Int J Chron Obstruct Pulmon Dis. 2008;3(2):285-93. doi: 10.2147/copd.s2654. PMID 18686737
- [Result] McClernon FJ, Westman EC, Rose JE. The effects of controlled deep breathing on smoking withdrawal symptoms in dependent smokers. Addict Behav. 2004 Jun;29(4):765-72. doi: 10.1016/j.addbeh.2004.02.005. PMID 15135559
- [Result] Tharion E, Samuel P, Rajalakshmi R, Gnanasenthil G, Subramanian RK. Influence of deep breathing exercise on spontaneous respiratory rate and heart rate variability: a randomised controlled trial in healthy subjects. Indian J Physiol Pharmacol. 2012 Jan-Mar;56(1):80-7. PMID 23029969
- [Result] Busch V, Magerl W, Kern U, Haas J, Hajak G, Eichhammer P. The effect of deep and slow breathing on pain perception, autonomic activity, and mood processing--an experimental study. Pain Med. 2012 Feb;13(2):215-28. doi: 10.1111/j.1526-4637.2011.01243.x. Epub 2011 Sep 21. PMID 21939499
- [Result] Shields RW Jr. Heart rate variability with deep breathing as a clinical test of cardiovagal function. Cleve Clin J Med. 2009 Apr;76 Suppl 2:S37-40. doi: 10.3949/ccjm.76.s2.08. PMID 19376980
- [Result] Song F, Holland R, Barton GR, Bachmann M, Blyth A, Maskrey V, Aveyard P, Sutton S, Leonardi-Bee J, Brandon TH. Self-help materials for the prevention of smoking relapse: study protocol for a randomized controlled trial. Trials. 2012 May 30;13:69. doi: 10.1186/1745-6215-13-69. PMID 22647290